CLINICAL TRIAL: NCT00801788
Title: Single Dose Pharmacokinetics of Egalet® Oxycodone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: OC-EG-001
Record Dates: First submitted 2008-12-02; First posted 2008-12-04 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Egalet® oxycodone Treatment A (Experimental): Single Dose Administration
  Interventions: Drug: Oxycodone hydrochloride
- Egalet® oxycodone Treatment B (Experimental): Single Dose Administration
  Interventions: Drug: Oxycodone hydrochloride
- Egalet® oxycodone Treatment C (Experimental): Single Dose Administration
  Interventions: Drug: Oxycodone hydrochloride
- Active comparator (Active Comparator): Single Dose Administration
  Interventions: Drug: Oxycodone hydrochloride

INTERVENTIONS:
Drug: Oxycodone hydrochloride — Extended release tablet
  Arms: Egalet® oxycodone Treatment A; Egalet® oxycodone Treatment B; Egalet® oxycodone Treatment C
Drug: Oxycodone hydrochloride — Extended release tablet
  Arms: Active comparator

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetic profile of different Egalet® oxycodone formulations and compare to a marketed oxycodone product.

ELIGIBILITY:
Main inclusion criteria:

* ≥18 years and ≤55 years
* Non-smoker
* BMI ≥18.0 and ≤30.0

Main exclusion criteria:

* Any clinically significant abnormality or abnormal laboratory test results found during medical screening
* History of allergic reactions to opioids or other related drugs
* History of significant alcohol abuse or drug abuse
* Use of any drugs known to inhibit hepatic drug metabolism
* Pregnant or breast-feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To evaluate pharmacokinetics of Egalet® oxycodone. AUC0-t, AUC0-inf, Cmax, Residual Area, Tmax, T½ el,Kel,AUC 0-12 and AUC 0-24. | Single-dose evaluation

SECONDARY OUTCOMES:
To evaluate safety and tolerability of Egalet® oxycodone. Hematology, biochemistry, urinalysis, vital signs (including pulse oximetry), and adverse event monitoring. | Single-dose evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Christine Andersen, M.Sc., Study Director — Egalet A/S
Locations (1):
- Québec, Quebec, Canada